CLINICAL TRIAL: NCT05021536
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of AMX0035 Versus Placebo for 48-week Treatment of Adult Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Phase III Trial of AMX0035 for Amyotrophic Lateral Sclerosis Treatment
Acronym: Phoenix
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A35-004
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — sodium phenylbutyrate and taurursodiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered by mouth or via feeding tube for 48 weeks: once daily for first 3 weeks and then twice daily for remainder of study if participant tolerating
  Interventions: Other: Placebo
- AMX0035 (Experimental): Placebo administered by mouth or via feeding tube for 48 weeks: once daily for first 3 weeks and then twice daily for remainder of study if participant tolerating
  Interventions: Drug: AMX0035

INTERVENTIONS:
Other: Placebo — Matching Placebo Comparator
  Arms: Placebo
Drug: AMX0035 — Proprietary formulation of taurursodiol and sodium phenylbutyrate
  Arms: AMX0035

SUMMARY:
The Phoenix Trial is a randomized double blind placebo controlled Phase III trial to evaluate the safety and efficacy of AMX0035 for treatment of ALS

DETAILED DESCRIPTION:
AMX0035 is a combination therapy designed to reduce neuronal death through blockade of key cellular death pathways originating in the mitochondria and endoplasmic reticulum (ER). This clinical trial is designed to demonstrate that treatment is safe, tolerable, and able to slow decline in function as measured by the ALSFRS-R and survival over 48 week. The trial will also assess the effects of AMX0035 on slow vital capacity, quality of life and plasma biomarkers of ALS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* Diagnosis of ALS (definite or clinically probable)
* Time since onset of first symptom of ALS should be <24 months prior to randomization;
* If the participant is to be treated with riluzole and/or edaravone during the course of the trial, then treatment with riluzole and/or edaravone was, at the time of the screening visit, started and maintained at a stable regimen for at least 14 days for riluzole and/or for a full treatment cycle for edaravone;
* Capable of providing informed consent
* Capable and willing to follow trial procedures including visits to the trial clinic and visit requirements;
* Women of child bearing potential (e.g. not post-menopausal for at least one year or surgically sterile) must agree to use adequate birth control for the duration of the study and 3 months after last dose of study drug. Women must not be planning to become pregnant for the duration of the study and 3 months after last dose of study drug
* Men must agree to practice contraception for the duration of the study and 3 months after last dose of study drug. Men must not plan to father a child or provide for sperm donation for the duration of the study and 3 months after last dose of study drug

Exclusion Criteria:

* Presence of tracheostomy or permanent assisted ventilation(PAV)
* Slow Vital Capacity (SVC) less than 55%
* History of known allergy to phenyl butyrate or bile salts
* Abnormal liver function defined as bilirubin levels and/or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 5 times the upper limit of the normal (obtained within 12 weeks from first dose)
* Renal insufficiency as defined by eGFR <60 mL/min/1.73m^2 (obtained within 12 weeks from first dose)
* Pregnant women (confirmed by a pregnancy test within 7 days of first dose) or women currently breastfeeding
* Current severe biliary disease which may result in the Investigator medical judgement in biliary obstruction including for example active cholecystitis, primary biliary cirrhosis, sclerosing cholangitis, gallbladder cancer, gangrene of the gallbladder, abscess of the gallbladder
* History of Class III/IV heart failure (per New York Heart Association - NYHA)
* Participant under severe salt restriction where the added salt intake due to treatment would put the participant at risk, in the Investigator clinical judgment
* Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that would impair ability of the participant to provide informed consent, according to Investigator judgment
* Clinically significant unstable medical condition (other than ALS) (e.g., cardiovascular instability, systemic infection, untreated thyroid dysfunction, severe laboratory test anomaly or clinically significant electrocardiogram [ECG] changes) that would pose a risk to the participant if he/she were to participate in the trial, according to Investigator judgment
* Previous treatment for ALS with cellular therapies or gene therapies
* Currently enrolled in another trial involving use of an investigational therapy
* Previous treatment with PB or taurursodiol within 30 days from Screening
* Implantation of Diaphragm Pacing System (DPS)
* Currently or previously treated within the last 30 days or planned exposure to any prohibited medications listed in Section 6.8 of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Slope Change | 48 weeks
  Change in slope of Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) over treatment duration. The ALSFRS-R consists of 12 items across 4 subdomains of function (bulbar, fine motor, gross motor, and breathing) with each item scored on a scale from 0 (total loss of function) to 4 (no loss of function). Total scores range from 0 to 48, with higher scores indicating better function.

SECONDARY OUTCOMES:
Participant Quality of Life (QOL) | 48 weeks
  QOL will be measured using the 40-item Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) patient-reported outcome (PRO)
Assess Long-Term Survival | 3 years from LPI
  Long-Term Survival will be obtained by monitoring of all-cause mortality
Rate of Decline in Slow Vital Capacity (SVC) | 48 weeks
  Respiratory muscle function will be assessed according to slow vital capacity (SVC). SVC is measured in an upright position for at least three trials per assessment. SVC volumes will be standardized to the percentage of predicted normal value based on age, sex, and height.
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Slope Change | 24 weeks
  Change in slope of Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) over treatment duration. The ALSFRS-R consists of 12 items across 4 subdomains of function (bulbar, fine motor, gross motor, and breathing) with each item scored on a scale from 0 (total loss of function) to 4 (no loss of function). Total scores range from 0 to 48, with higher scores indicating better function.
Number of Participants With Adverse Events | 48 weeks
  Comparison Between Groups of Number of Participants With Adverse Events Until Planned Completion

CONTACTS AND LOCATIONS:
Overall Officials: Amylyx Study Director, Study Director — Amylyx Pharmaceuticals
Locations (69):
- United States (28):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - University of California Irvine, Orange, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University Neuroscience Center, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University School of Medicine Outpatient Center, Baltimore, Maryland
  - Healey & AMG Center for ALS Research at Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - Rutgers University, New Brunswick, New Jersey
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
  - Texas Neurology, Dallas, Texas
  - Virginia Commonwealth University, Henrico, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - University of Washington, Seattle, Washington
- University Hospitals Leuven, Leuven, Belgium
- France (9):
  - Hospices Civils de Lyon Hôpital Neurologique Pierre Wertheimer Cellule Mutualisée de Recherche Clinique (CMRC), Bron
  - Hopital Gabriel Montpied Service de Neurologie, Clermont-Ferrand
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hôpitaux Universitaires de Marseille Timone, Marseille
  - CHU de Montpellier, Montpellier
  - CHU Nice, Nice
  - Hôpital de la Salpêtrière, Paris
  - Le Centre Hospitalier Régional Universitaire de Tours, Tours
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Uniklinikum Dresden, Dresden
  - Hannover Medical School, Hanover
  - Jena University Hospital, Jena
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
  - University Medical Center Rostock, Rostock
  - Ulm University Medical Centre, Ulm
- Trinity College Dublin/Beaumont Hospital, Dublin, Ireland
- Italy (7):
  - Università degli Studi di Bari Aldo Moro, Bari
  - Centro Clinico NEMO, Milan
  - University of Milan Medical School, Milan
  - Azienda Ospedaliero Universitaria Di Modena, Modena
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - University of Padua, Padua
  - University of Torino, Turin
- University Medical Center Utrecht, Utrecht, Netherlands
- Poland (2):
  - Centrum Medyczne Linden, Krakow
  - City Clinic Warsaw, Warsaw
- Centro Hospitalar Universitário Lisboa-Norte, Lisbon, Portugal
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital Universitari de Bellvitge-IDIBELL, Barcelona
  - Hospital San Rafael, Madrid
  - Biodonostia Health Research Institute; Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario y Politécnico La Fe, Valencia
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Umeå University Hospital, Umeå
- United Kingdom (5):
  - King's College London, London
  - UCL Queen Square Institute of Neurology, London
  - University of Plymouth, Plymouth
  - Salford Royal Hospital Barnes, Salford
  - Sheffield Institute for Translational Neuroscience (SITraN), Sheffield